CLINICAL TRIAL: NCT00995332
Title: Treatment of Acute Myelogenous Leukemia With the Histone Deacetylase Inhibitor Valproic Cid in Combination With All-trans Retinoic Acid (ATRA) and Low Dose Cytarabine
Brief Title: Disease Stabilization in AML by Treatment With ATRA, Valproic Acid and Low-dose Cytarabine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Øystein Bruserud, Professor, University of Bergen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rek VEST 231-06
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute myelogenous leukemia; all-trans retinoic acid; valproic acid; cytarabine; Disease stabilization; survival; toxicity
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Tretinoin; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATRA+valproc acid+low-dose cytarabine (Experimental)
  Interventions: Drug: Cytarabine, all-trans retinoic acid, valproic acid

INTERVENTIONS:
Drug: Cytarabine, all-trans retinoic acid, valproic acid — ATRA: 22.5 mg/m2 twice daily for 2 weeks every third month Valproic acid: continuous therapy, dosage guided by serum levels Cytarabine: 10 mg/m2 once daily for up to 10 days every third month
  Other Names: No other names

SUMMARY:
Hypothesis: Combined treatment with valproic acid and ATRA can be used to achieve disease stabilization for a subset of patients with acute myelogenous leukemia (AML), and this effect can be improved without serious toxicity by adding low-dose cytarabine to this treatment.

Adult patients >18 years of age who can be included:

Elderly patients who cannot achieve standard chemotherapy, patients with relapsed or resistant AML.

Treatment: Combined therapy with:

Valproic acid, continuous therapy until disease progression ATRA, oral therapy for 14 days every three months Low-dose cytarabine 10 mg/m2 up to 10 injections during week 2 and 3, repeated every 3 months.

DETAILED DESCRIPTION:
Patients to be included:

1. Elderly patients (>60 years of age) or other patients unfit for conventional intensive chemotherapy with newly diagnosed acute myelogenous leukemia (AML).
2. Adult patients of any age (>18 years of age) with relapsed or resistant AML who cannot receive conventional therapy.

Treatment:

Valproic acid to be started on day 1 as continuous therapy until disease progression.

ATRA administered from day 8 orally as 22.5 mg/m2 twice daily for 14 days, repeated every third month.

Low-dose cytarabine 10 mg/m2 from day 14 and continued as daily injections for up to 10 days, repeated every third month.

Supportive therapy is given according to the hospitals general guidelines.

Followup: The first 2 days treatment in hospital, later regular out-patient treatment. Controls will include clinical examination, peripheral blood parameters (including serum valproic acid levels), bone marrow samples.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed AML in patients unfit for intensive chemotherapy
* Patients with relapsed or refractory AML

Exclusion Criteria:

* No informed consent
* Intolerance to study drugs
* Serious liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Survival | 3 years

SECONDARY OUTCOMES:
Disease stabilization | 3 years
Disease complications | 3 years
Side effects of therapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Oystein Bruserud, MD, Study Chair — University of Bergen, Norway
Locations (1):
- Haukeland University Hospital and University of Bergen, Bergen, Norway

REFERENCES:
- [Background] Fredly H, Ersvaer E, Kittang AO, Tsykunova G, Gjertsen BT, Bruserud O. The combination of valproic acid, all-trans retinoic acid and low-dose cytarabine as disease-stabilizing treatment in acute myeloid leukemia. Clin Epigenetics. 2013 Aug 1;5(1):13. doi: 10.1186/1868-7083-5-13. PMID 23915396
- [Derived] Haaland I, Hjelle SM, Reikvam H, Sulen A, Ryningen A, McCormack E, Bruserud O, Gjertsen BT. p53 Protein Isoform Profiles in AML: Correlation with Distinct Differentiation Stages and Response to Epigenetic Differentiation Therapy. Cells. 2021 Apr 7;10(4):833. doi: 10.3390/cells10040833. PMID 33917201
- [Derived] Reikvam H, Hovland R, Forthun RB, Erdal S, Gjertsen BT, Fredly H, Bruserud O. Disease-stabilizing treatment based on all-trans retinoic acid and valproic acid in acute myeloid leukemia - identification of responders by gene expression profiling of pretreatment leukemic cells. BMC Cancer. 2017 Sep 6;17(1):630. doi: 10.1186/s12885-017-3620-y. PMID 28877686